CLINICAL TRIAL: NCT06240533
Title: Implementation of a Patient Centered Coordinated Care Pathway for Low Back Pain (P3C-LBP) in Swedish Primary Care
Brief Title: Implementation of P3C-LBP in Swedish Primary Care
Acronym: P3C-LBP
Status: Not yet recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Allan Abbott, Professor, Linkoeping University
Other Study IDs: 20240201
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: Implementation; Care pathway; Patient centered care; Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Historical baseline: Patients with LBP in a retrospective register based study of health care quality indicators covering historical time series data from regional health care databases in Sweden before dissemination by publication of the P3C pathway (January 2013-June 2023).
- Dissemination: Patients with LBP in a prospective register based study of health care quality indicators for phase 1 (January 2013-June 2023) compared to phase 2 (June 2023- February 2024) after dissemination by publication of the P3C pathway for LBP.
- Single-faceted implementation: Patients with LBP in a prospective register based study of health care quality indicators for phases 1+2 (January 2013-February 2024) compared to phase 3 (March 2024-February 2026) after single-faceted implementation (health care practitioner workshop) of the P3C pathway for LBP. Health care practitioner confidence in managing LBP and perspectives regarding barriers and facilitators determining implementation P3C pathway success will also be investigated via questionnaires and qualitative interviews directly after and 1 year prospectively the implementation intervention.
- Multi-faceted implementation: Patients with LBP in a prospective register based study of health care quality indicators for phases 1+2+3 (January 2013-February 2026) compared to phase 4 (March 2026-December 2027) after multi-faceted implementation (repeated health care practitioner workshops and follow-up) of the P3C pathway for LBP.

SUMMARY:
The goal of this observational study is to evaluate the implementation of a patient centered coordination care (P3C) pathway for the management of patients with low back pain (LBP) in primary care, in Östergötland health care region, Sweden.

The main questions the study aims to answer are:

* Do health care quality indicators improve over time after repeated implementation interventions of a P3C pathway for patients with LBP.
* What are the health care practitioner perspectives regarding barriers and facilitators determining implementation success of a P3C pathway for patients with LBP.

DETAILED DESCRIPTION:
BACKGROUND Since 2019, the Swedish government together with regional health care organisations have actioned the national development of patient centered coordinated care (P3C) pathways. P3C pathways are defined as health care processes guided by and organized effectively around the needs and preferences of the patient. The aim of this observational study is to evaluate the implementation of a patient centered coordination care (P3C) pathway for the management of patients with low back pain (LBP) in primary care, Östergötland health care region, Sweden. The P3C pathway covers primary care processes until the patient can self-manage or transitions to established chronic pain or other specialist care pathways. A national work group was formed consisting of representatives from all regional health care organisations in Sweden and included all relevant health care professions, academia, and patient organisations.

METHODS:

A mixed methods iterative design and consensus approach was applied in the development of the P3C pathway. The study will be performed in 3 phases:

Phase 1 - Historical baseline: Retrospective register based study of health care quality indicators covering historical time series data before dissemination of the P3C pathway for LBP (January 2013-June 2023).

Phase 2 - Dissemination by publication: Prospective register based study of health care quality indicators for phase 1 (January 2013-June 2023) compared to phase 2 (June 2023- February 2024) after dissemination by publication of the P3C pathway for LBP.

Phase 3 - Single-faceted implementation: Prospective register based study of health care quality indicators for phases 1+2 (January 2013-February 2024) compared to phase 3 (March 2024-February 2026) after single-faceted implementation (health care practitioner workshop) of the P3C pathway for LBP. Health care practitioner confidence in managing LBP and perspectives regarding barriers and facilitators determining implementation P3C pathway success will also be investigated via questionnaires directly after and 1 year prospectively after the implementation intervention. The qualitative interviews will be performed 3- 6 months post implementation.

Phase 4 - Multi-faceted implementation (repeated health care practitioner workshops and follow-up): Prospective register based study of health care quality indicators for phases 1+2+3 (January 2013-February 2026) compared to phase 4 (March 2026-December 2027) after multi-faceted implementation of the P3C pathway for LBP.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with the low back diagnosis (M.54.5, M54.4, M54.3, M54.9) with a visit in primary care and patients with diagnosis M43.0,M43.1, M43.9,M47(all but not M47.0),M48.0, M48.0K, M48.8,M48.8K, M48.9, M51.0, M51.0K, M51.1,M51.1K, M51.2, M51.3, M51.4, M51.8, M51.9, M53.2, M53.3, M53.8,M53.9 referred from primary to specialist care for LBP.
2. General practitioners and primary health care nurses participating in P3C implementation workshops

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population for outcomes 2,3&6-15 is patients with low back pain seeking primary care for low back pain between 2013 to 2027
  Study population for outcome 1,4,5 is General practitioners and nurses in primary care in the region of Östergötland who attend the implementation workshop education during February 2024.
  Study population for outcome 4 is General partitioners and nurses in primary care in the region of Östergötland who have not attended the implementation education workshop and are willing to participate in an interview during May to october 2024.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Practitioner Confidence Scale | February 2024 and February 2025
  Healthcare practitioner rated´confidence in managing low back pain before and after a single-faceted implementation. The Practitioner Confidence Scale contains four items reported on a 5-point Likert scale, where a total score of 4 represents greatest self-confidence and 20 represents lowest self-confidence for managing patients with LBP.
Patient sickness benefit days per month for LBP | Monthly January 2013 to December 2027
  Registry data from The Swedish Social Insurance Agency for diagnosis codes (ICD10: M54.5, M54.4, M54.3, M54.9)
Cost of health care per month for LBP | Monthly January 2013 to December 2027
  Registry data from the Östergötland health care region database for diagnosis codes (ICD10: M54.5, M54.4, M54.3, M54.9)

SECONDARY OUTCOMES:
Determinants of Implementation Behaviour Questionnaire | February 2024 and February 2025
  Healthcare practitioners self rated barriers and facilitators determining implementation of the P3C pathway for LBP. Contains 10 items with 9-point Likert response scales ranging from 1='totally agree' to 9='totally disagree'.
Qualitative focus group interview | September 2024 to May 2025
  Healthcare practitioners´ will be interviewed to explore barriers and facilitators determing the implementation of the P3C pathway for LBP
Use of medical imaging for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (ICD10: M54.5, M54.4, M54.3, M54.9) who have been investigated by medical imaging (KVÅ codes AN022, AN023, AN024; AN025, AN026, AN044, AN045, AN065, AN067, AN068).
Prescription of NSAIDS for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M54.5, M54.4, M54.3, M54.9) who have been prescribed the following drugs ATC prescription codes for NSAIDS (M01AB01, M01AB02, M01AB05, M01AB55, M01AC01, M01AC02, M01AC05, M01AC06, M01AE01, M01AE02, M01AE03, M01AE14, M01AE52, N02BA01, N02BA51, N02BB01, N02BB51, M02AA10, M02AA13, M02AA15, M01AH01, M01AH05, M01AH06, M01AX01)
Prescriptions of paracetamol for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M54.5, M54.4, M54.3, M54.9) who have been prescribed the following drugs ATC prescription codes for paracetamol (N02BE01, N02BE51).
Prescriptions of opioids for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M54.5, M54.4, M54.3, M54.9) who have been prescribed the following drugs ATC prescription codes for opioids (N02AA59, N02AC04, N02AE01, N02AJ06, N02AJ08, N02AJ09, N02AX02, N02AX06, N02AA01, N02AA03, N02AA05, N02AA55, N02AB01 N02AB03, N02AG01, N02AG02)
Prescriptions of gabapentinoids for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M54.4, M54.3, M48.0K, M48.8K, M51.0, M51.0K, M51.1, M51.1K) who have been prescribed the following drugs ATC prescription codes for gabapentinoids (N03AX12, N03AX16, N02BF01, N02BF02)
Prescriptions of antidepressants for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M54.4, M54.3, M48.0K, M48.8K, M51.0, M51.0K, M51.1, M51.1K) who have been prescribed the following drugs ATC prescription codes for antidepressants (N06AX21, N06AB05, N06AB03, N06AA02, N06AA09, N06AA12, N06AA10, N06AA01, N06AX12, N06AX17)
Prescriptions of muscle relaxants for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M54.5, M54.4, M54.3, M54.9) who have been prescribed the following drugs ATC prescription codes for muscle relaxant drugs (M03BB03, M03BC51, M03BA02, M03BX08, M03BX05, N04AB02, M03BA03, M03BX01, N05BA01)
Referrals to specialist orthopedic clinics | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M43.0, M43.1, M43.9, M47(all except M47.0), M48.0, M48.0K, M48.8, M48.8K, M48.9, M51.0, M51.0K, M51.1, M51.1K, M51.2, M51.3, M51.4, M51.8, M51.9, M53.2, M53.3, M53.8, M53.9) who have been referred to specialized care - orthopaedic clinic.
Referrals to specialist pain rehabilitation clinics | Monthly January 2013 to December 2027
  Number of patients per month with new visits to primary care due to diagnosis codes (M43.0, M43.1, M43.9, M47(all except M47.0), M48.0, M48.0K, M48.8, M48.8K, M48.9, M51.0, M51.0K, M51.1, M51.1K, M51.2, M51.3, M51.4, M51.8, M51.9, M53.2, M53.3, M53.8, M53.9) who have been referred to specialist care - pain rehabilitation clinics.
New visits in primary care to physicians and physiotherapists for LBP | Monthly January 2013 to December 2027
  Number of patients per month with new visits to physicians and number of patients per month with new visits to physiotherapists in primary care due to diagnosis codes (M54.5, M54.4, M54.3, M54.9).

CONTACTS AND LOCATIONS:
Overall Officials: Allan Abbott, Professor, Principal Investigator — Department of Health, Medicine and Caring Sciences, Linköping University, Sweden; Allan Abbott, Professor, Study Chair — Department of Health, Medicine and Caring Sciences, Linköping University, Sweden; Allan Abbott, Professor, Study Director — Department of Health, Medicine and Caring Sciences, Linköping University, Sweden
Locations (1):
- Östergötland health care region, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Registry data is owned by the Swedish government